CLINICAL TRIAL: NCT00037531
Title: An Open-label Extension Study of the Safety of Long-term Administration of Sirolimus (Rapamune™) in Solid Organ Transplant Recipients
Brief Title: Study Evaluating Sirolimus (Rapamune™) in Solid Organ Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 0468E1-306
Record Dates: First submitted 2002-05-17; First posted 2002-05-20 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Graft vs Host Disease; Kidney Transplantation
Keywords: Transplant; Kidney
MeSH Terms: conditions — Graft vs Host Disease | interventions — Sirolimus

INTERVENTIONS:
Drug: Sirolimus (RAPAMUNE)

SUMMARY:
To evaluate the safety of long-term administration of sirolimus oral solution for up to 5 additional years, or until the tablet formulation is commercially available (whichever occurs first) in solid organ transplant recipients who are currently receiving sirolimus and who have completed clinical trials with sirolimus (with or without cyclosporine (CsA). To evaluate the pharmacokinetics and safety of long-term administration of sirolimus tablets administered for up to 5 years, or until the tablet formulation is commercially available in solid organ transplant recipients who are currently receiving sirolimus and who have completed clinical trials with sirolimus (with or without CsA) or who are currently enrolled in protocol 0468E1-306-US.

ELIGIBILITY:
Inclusion Criteria:

* Completion of sirolimus/blinded therapy in solid organ clinical trials (with or without CsA) with satisfactory compliance and an adequate safety profile.
* Women of childbearing potential who have a negative pregnancy test before enrollment into this study and who agree to practice either a hormonal or barrier method of birth control throughout the treatment period and for 3 months following discontinuation of sirolimus may be enrolled into the study.
* Signed and dated informed consent

Exclusion Criteria:

* Unstable disease states, which in the opinion of the investigator would present a risk to the patient.
* Known hypersensitivity to macrolide antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 769 (Actual)
Dates: Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (18):
- United States (13):
  - Los Angeles, California
  - San Diego, California
  - Stanford, California
  - Tampa, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - New York, New York
  - Charlotte, North Carolina
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
- Canada (5):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - Toronto, Ontario
  - Montreal, Quebec